CLINICAL TRIAL: NCT05183893
Title: Malate or Not?: Effects of L-Citrulline or Citrulline-malate on Neuromuscular Performance in Resistance-trained Adults
Brief Title: Effects of L-Citrulline or Citrulline-malate on Neuromuscular Performance in Resistance-trained Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Lucas Jurado-Fasoli, Researcher, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: Malate or Not Project
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Neuromuscular Performance
Keywords: nitric oxide; dietary supplement; resistance training; citrulline malate
MeSH Terms: interventions — Citrulline; citrulline malate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: L-Citrulline (Experimental): 5 g of L-citruline + 5 g of additives. The dose to be administered is that recommended on the labeling and nutritional information of the product, which has been produced under GMP procedures and approved by the EFSA (Lifepro®).
  Interventions: Dietary Supplement: L-citrulline
- Experimental: Citrulline-malate (Experimental): 8g of citrulline-malate + 2 g of additives. The dose to be administered is that recommended on the labeling and nutritional information of the products which has been produced under GMP procedures and approved by the EFSA (Lifepro®).
  Interventions: Dietary Supplement: Citrulline-malate
- Placebo (Placebo Comparator): 10g of maltodextrin plus additives (Lifepro®).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-citrulline — 5 g of L-citruline + 5 g of additives
  Arms: Experimental: L-Citrulline
Dietary Supplement: Citrulline-malate — 8g of citrulline-malate + 2 g of additives
  Arms: Experimental: Citrulline-malate
Dietary Supplement: Placebo — 10g of maltodextrine
  Arms: Placebo

SUMMARY:
The main aim of this study is to compare the effects of L-Citrulline vs. Citrulline-malate on neuromuscular performance (maximal dynamic strength and maximal endurance strength) in resistance-trained adults.

DETAILED DESCRIPTION:
Nitric oxide (NO) is a ubiquitous gaseous molecule that plays a critical role in the regulation of cardiovascular function and in the signaling of multiple cellular processes. Specifically, NO could reduce the oxygen cost of exercise and adenosine triphosphate (ATP) in the production of muscle contractile force, improving calcium handling, glucose uptake and mitochondrial efficiency in muscle fibers. Therefore, it has been suggested that increasing the availability of NO through the oral intake of food and nutritional supplements may be useful to delay the onset of fatigue and improve performance in high-intensity efforts.

L-citrulline is a nonessential amino acid involved in the urea cycle that acts as an endogenous precursor of L-arginine, being a more efficient alternative to L-arginine to increase the plasma concentration of L-arginine through the nitric oxide synthase (NOS) pathway.

On the other hand, citrulline malate is an organic salt of L-citrulline and malate which has been shown to exert a small but significant ergogenic effect in different high-intensity efforts compared to a placebo. However, no study to date has compared L-citrulline VS. citrulline malate to assess whether there is an additive effect from malate to exercise performance.

50 resistance-trained adults (50% women) will be randomized into three conditions (L-citrulline, citrulline-malate and placebo conditions) with 48 hours of separation between conditions. 48h previous to the randomization the participants will perform a familiarization to avoid the learning effects.

Each evaluation day will conform to the following tests:

* Maximal dynamic strength of lower- and upper-body
* Maximal endurance strength of lower- and upper-body

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-30years
* BMI: 18-30.0 kg/m2
* Stable weight over the last 3 months (body weight changes<3kg)
* Previous experience in resistance training (i.e., at least 1 year with a frequency of two or more training sessions per week),
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols.

Exclusion Criteria:

* History of chronic diseases (renal disease, diabetes, cardiovascular disease, cancer, VIH, hepatic disease, food disorders)
* Pregnant, planning to become pregnant, or breastfeeding
* Have been treated previously or during the study period with prescription drugs:

antihypertensive, lipid lowering, acid uric lowering, glucose lowering, beta blockers or any drug that under the investigator's judged could influence the results.

* Allergy/intolerance to any ingredient of the dietary supplements.
* Chronic consumers of dietary NO-precursors dietary supplements (citrulline malate, arginine, nitrates).
* Any non-controlled medical condition which could influence results or could be worsened by the participation in the study.
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Maximal endurance strength | 1 hour
  Maximal endurance strength of lower- and upper-body (squat and bench press exercises)

SECONDARY OUTCOMES:
Maximal dynamic strength | 1 hour
  Maximal dynamic strength of lower- and upper-body (squat and bench press exercises)

CONTACTS AND LOCATIONS:
Locations (1):
- Jonatan Ruiz Ruiz, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martin-Olmedo JJ, Miras-Moreno S, Cuadra-Montes K, Garcia-Ramos A, Ruiz JR, Jurado-Fasoli L. Malate or Not? Acute Effects of L-Citrulline Versus Citrulline Malate on Neuromuscular Performance in Young, Trained Adults: A Randomized, Double-Blind, Placebo-Controlled Crossover Trial. Int J Sport Nutr Exerc Metab. 2024 Dec 11;35(2):89-98. doi: 10.1123/ijsnem.2024-0006. Print 2025 Mar 1. PMID 39662304